CLINICAL TRIAL: NCT04749862
Title: Patient Centred Models for Surveillance and Support of Cancer Survivors with Breast and Bowel Cancer
Brief Title: Cancer Surveillance and Support
Acronym: CANVAS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor, University of Leeds
Other Study IDs: L424
Record Dates: First submitted 2021-01-11; First posted 2021-02-11 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Breast Cancer Participants-Before Phase: Breast cancer patients (16 years old or over) who have completed active treatment will complete a series of patient reported outcomes at baseline, 3, 6 and 12 months time.
- Colorectal (bowel) Cancer Participants-Before Phase: Colorectal cancer patients (16 years old or over) who have completed active treatment will complete a series of patient reported outcomes at baseline, 3, 6 and 12 months time.
- Breast Cancer Participants-After Phase: Breast cancer patients (16 years old or over) who have completed active treatment will complete a series of patient reported outcomes at baseline, 3, 6 and 12 months time. In addition they will also complete an online symptom report from home with self-management advice (frequency of completion to be determined in phase 2)
  Interventions: Other: Online symptom reporting
- Colorectal (bowel) Cancer Participants-After Phase: Colorectal cancer patients (16 years old or over) who have completed active treatment will complete a series of patient reported outcomes at baseline, 3, 6 and 12 months time. In addition they will also complete an online symptom report from home with self-management advice (frequency of completion to be determined in phase 2)
  Interventions: Other: Online symptom reporting

INTERVENTIONS:
Other: Online symptom reporting — Online symptom reporting questionnaire with linked self-management advice
  Groups: Breast Cancer Participants-After Phase; Colorectal (bowel) Cancer Participants-After Phase

SUMMARY:
This project aims to enhance the support for patients with breast and bowel cancer after treatment. Current follow-up care includes either self-management with patient-initiated contacts (breast cancer) or scheduled hospital visits for scans/tests for recurrence (bowel cancer). Building on extensive experience with online patient self-reporting of symptoms during treatment, the study will develop, implement and evaluate satisfaction with an improved electronic system to engage breast and bowel cancer survivors to self-report symptoms/problems online from home and get immediate tailored advice for self-management or hospital contact. The reports are displayed real-time in the hospital records alongside scans/tests to inform clinical management.

DETAILED DESCRIPTION:
A structured plan of development, evaluation and implementation is proposed, based on the Medical Research Council (MRC) complex interventions framework and the principles of Action Research model (namely; Purpose choice on solving practical problems; Contextual focus; Data that helps track changes and sense making; Participation in research process and Knowledge diffusion). Action research is suited to identifying problems in clinical practice and helping develop potential solutions in order to improve practice. The study will use an experimental action research approach incorporating the action research cycle (Plan Do Study Act).

The effectiveness evaluation of patient/clinician acceptance, feasibility, patient benefits/satisfaction will be performed using a non-randomised 'Before-After study' approach, followed by immediate implementation in practice for faster patient benefits.

Main outcomes measured will include:

1. Patient-Reported Outcomes questionnaires: quality of life, symptom control, and self-efficacy.
2. Clinical measures: number of hospital contacts, recurrence rates.
3. Process measures: survivors compliance with self-reports, clinical tests attendance; using online self-management resources.

The project will be structured in four phases:

PHASE 1 (Months 0-12): Develop the content of the surveillance toolkits for breast and bowel (colorectal) cancers and setup on the electronic system. This will include the selection of cancer-specific symptoms for patient self-reporting, collating the existing evidence on side-effects management and the development of patient advice corresponding to severity levels. Once the two toolkits for breast and bowel (colorectal) cancers are completed, they will be set up on the electronic system. Printed booklets can also be produced from these.

Recruitment methods:

Cancer survivors and caregivers will be invited from outpatient surveillance clinics or by telephone by the cancer team if discharged recently from secondary care, and by public advertising for breast and colorectal cancer survivors volunteers. Purposive sampling will represent a variety of age groups, cancer recurrence risk, time post treatment, socio-economic background, expecting a sample of 8-10 survivors/carers per cancer site. Participants will be invited for an interview conducted over the telephone or at St James's Hospital.

Healthcare professionals (HCP) involved in breast and colorectal cancer care at St James's Hospital will also be invited to participate in interviews. This is done face to face at the hospital followed up by a phone call or an individual email depending on the previous conversations had between the researchers and the HCP.

Interviews will be transcribed verbatim and subjected to thematic content analysis.

Phase 1 Objectives:

1. Select questions for self-reporting
2. Determine severity thresholds
3. Determine content of the self-management guidance
4. Describe the current usual care after treatment by cancer type and how to modify it to incorporate remote surveillance
5. Identify potential improvements to the electronic system.

PHASE 2:"Before study" (Months 6-30; 12-months recruitment,12-months follow-up)The before study will be a structured audit of current practice, running in parallel with Phase 1.

Participants who consent will complete outcome measures at baseline, 3, 6 and 2 months on paper. Demographic data will be collected after consent and clinical data will be collected via the EPR.

Recruitment methods:

The study will include recruitment over 12 months of all consecutive eligible patients with a follow-up of 12 months. The estimated numbers are 120 new bowel (colorectal) cancer patients per year and 300 breast cancer patients. The study anticipates 70% consent rate, giving approximately 85 bowel (colorectal) and 210 breast cancer participants.

Phase 2 Objectives:

1. Establish data on current practice using clinical and patient outcomes and best methods for collecting them
2. Provide 'Before' data to compare to "After study" to estimate the effects of the new intervention
3. Establish prospectively what proportion of eligible patients would consent to a remote monitoring study.

PHASE 3:"After study"(Months 18-42;12-months recruitment, 12-months follow-up) Participants will be completing the intervention for 12 months. The 'After study' will start when Phase 1 is completed, including a successful usability testing.

Participants who consent will complete outcomes measures at baseline, 3, 6 and 12 months on paper (same as Phase 2). In addition, they will also complete the intervention: online symptom reporting questionnaire.

Demographic data will be collected after consent and clinical data via the Electronic patient records (EPR).

Recruitment methods:

Based on current experience of other studies conducted 15% of breast and 20% of bowel (colorectal) patients will not use online resources. Therefore, the estimated number of full participants will be about 170 in breast and 70 in bowel (colorectal) cancer clinics. The remote monitoring will only be available to participants classed as being moderate to lower risk by their clinical team. The intervention is an additional service for patients conducted along side their standard cancer care.

Phase 3 Objectives:

1. Assess the effects of the intervention in terms of participants' quality of life at baseline, 3, 6 and 12 months
2. Examine survivors' engagement with the intervention - acceptability, feasibility and use of the online system and respective advice
3. Examine clinicians' engagement

   Secondary objectives:
4. Monitor the safety i.e. diagnoses of recurrences and psychological morbidity, how were those detected
5. Evaluate impact on participants' self-efficacy in managing cancer consequences and fear of recurrence
6. Evaluate participants' satisfaction with care
7. Compare use of National Health Service (NHS) resources in Before and After phase.

The implementation of the intervention:

The intervention (as developed in Phase 1) will be implemented following the relevant staff and participant training. The frequency of participants' completions will be determined in Phase 1. Participants will be asked to complete the online symptom monitoring from home, with the possibility to complete the questions more often, if they experience any symptoms they may wish to report. Text message or email reminders will be sent to the participants (based on their preferred contact method) as a prompt to complete the online monitoring symptom questions, and where relevant to attend for the blood tests or surveillance scans.

Providers are expected to review and respond to any notifications for significant symptoms, in line with the agreed thresholds and are expected to review the self-reports during the clinic visits, discuss them with the patient and take any actions, as appropriate.

Participants and staff interviews will be conducted during and at the end of Phase 3.

PHASE 4: (starting month 30, with specific launch activities 42-48): Roll-out and implementation in practice. Following the principles of the Action research model (Act phase), the aim is to start roll-out immediately after completion of the 12-month recruitment in the "After" study. This will involve further work to apply the learning from Phase 3:

1. Simplify patient approach and consent to integrate it into the routine clinics flow
2. Identify appropriate clinic staff to approach patients
3. Modify, if needed, the self-reported questions, the thresholds or the content of the advice.

ELIGIBILITY:
Inclusion Criteria:

* Breast and colorectal healthcare professionals (e.g. Clinical Nurse Specialists) working at St James' University Hospital

Participating patients Phases 1 and 2:

* Patients (aged 16 years or over) attending St James' University Hospital Bexley Wing, with breast and/or colorectal cancer in remission, completed their cancer treatment.
* Able and willing to give informed consent
* Able to read and understand English

Participating patients Phase 3:

* Patients (aged 16 years or over) attending St James' University Hospital Bexley Wing, with breast and/or bowel (colorectal) cancer in remission, completed their cancer treatment.
* Able and willing to give informed consent
* Able to read and understand English
* Access to the internet

Exclusion Criteria:

* Patients under the age of 16
* Patients exhibiting overt psychopathology/cognitive dysfunction
* Patients taking part in other clinical trials involving the completion of extensive patient reported outcome or quality of life measures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast and Colorectal cancer patients who have completed active treatment (up to 12 months after end of treatment).
Sampling Method: Non-Probability Sample
Enrollment: 565 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life after cancer treatment | 2021-2023
  To assess the effects of the online intervention on participants' health related quality of life after cancer treatment for colorectal and breast.
  1. Quality of Life in Adult Cancer Survivors scale (QLACS): Questions rated on a 1-7 point response scale, ranging from "never" to "always".
Disease Specific Quality of Life after cancer treatment in Colorectal - EORTC QLQ-CR29 | 2021-2023
  1. European Organisation for Research and Treatment of Cancer: EORTC QLQ colorectal module respectively (CR29): Questions are rated on a 4-7 point scale and overall scale scores are calculated from 0-100 with higher scores indicating better quality of life.
Disease Specific Quality of Life after cancer treatment in Breast- EORTC QLQ-BR49 | 2021-2023
  1. European Organisation for Research and Treatment of Cancer: EORTC QLQ breast module respectively (BR49): Questions are rated on a 4-7 point scale and overall scale scores are calculated from 0-100 with higher scores indicating better quality of life.
Intervention engagement: participant withdrawals | 2022-2023
  To examine participants' engagement with the intervention.
  1) Number of participant withdrawals from the study.
Intervention engagement: participants returning to routine follow-up. | 2022-2023
  To examine participants' engagement with the intervention.
  1) Number of patients who moved back to routine follow-up (from remote follow-up).
Intervention engagement: Participants' views on the online system. | 2022-2023
  To examine participants' engagement with the intervention.
  1) Participants qualitative interviews.
Clinician engagement | 2022-2023
  To examine clinicians' engagement with the intervention. Clinician qualitative end of study interviews.
Participant Recruitment | 2021-2023
  Recruitment, follow-up and attrition.
  1. Number of potentially eligible patients, number approached, number recruited vs. number not recruited, reasons for ineligibility and reasons for non-consent.
  2. Comparison of patient characteristics in before and after phase.
  3. Number of withdrawals.

SECONDARY OUTCOMES:
Patient Safety | 2022-2023
  To monitor the safety i.e. diagnoses of recurrences.
  1) Time to recurrence/relapse and method of diagnosis (symptoms, tumour markers, scans) via Electronic patient records (EPR).
Patients' Self-efficacy in managing their cancer | 2021-2023
  To assess participants' self-efficacy in managing their cancer via a 6-item self-efficacy scale.
  1. Self-efficacy-Lorig 6-item scale. Questions are rated on a 1 to 10 point response scale, ranging from "not at all confident" to "totally confident".
National Health Service (NHS) Resources | 2021-2023
  To compare use of National Health Services (NHS) resources in the Before and the After phase.
  1) Use of resources by patients - via a tailored Health Economics questionnaire.
Intervention implementation process measures: participant adherence | 2022-2023
  Measures of implementation of the intervention.
  1) Measures of implementation of the intervention - participants' adherence to regular online reporting.
Intervention implementation process measures: frequency of reported problems | 2022-2023
  Measures of implementation of the intervention.
  1) Measures of implementation of the intervention - participants' frequency of self-reported problems and relevant advice provided.

OTHER OUTCOMES:
Information systems | 2022-2023
  To assess the integrity of the information systems.
  1) Number of problems/issues with using the integrated system recorded via phone calls/emails from participants or clinical users to the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No